CLINICAL TRIAL: NCT06159530
Title: Effect Of Occlusal Materials Used For All On Four Implant Supported Mandibular Fixed Prosthesis With PEEK Framework
Brief Title: Effect Of Occlusal Materials Used For All On Four Mandibular Implant Prosthesis With PEEK Framework
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed shady, Assistant Professor, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A03021121
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Occlusal Trauma
MeSH Terms: interventions — Dental Implants

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEEK framework veneered with nanocomposite resin(visio-lign) (Experimental): patients recieved 4 implants according to All on 4 concept then peek framework was delivered and veneered with nano-composite resin (visio-lign) as an occlusal material
  Interventions: Procedure: dental implants; Procedure: peek framework; Procedure: visio-lign nano composite
- PEEK framework veneered with zirconia crowns (Experimental): patients recieved 4 implants according to All on 4 concept then peek framework was delivered and veneered with zirconia crowns as an occlusal material
  Interventions: Procedure: dental implants; Procedure: peek framework; Procedure: zirconia crowns

INTERVENTIONS:
Procedure: dental implants — 4 dental implants placed in the mandible according to all-on 4 concept
Procedure: peek framework — peek framework screwed to multi-unit abutments of 4-implants
Procedure: visio-lign nano composite — peek framework veneered with nano composite (visio-lign) as an occlusal material
  Arms: PEEK framework veneered with nanocomposite resin(visio-lign)
Procedure: zirconia crowns — peek framework covered with zirconia crowns as an occlusal material
  Arms: PEEK framework veneered with zirconia crowns

SUMMARY:
This study was performed to compare between the effects of different occlusal materials used for all on four implant supported mandibular fixed prosthesis with PEEK framework.

Methods of Evaluation

1- Occlusal force analysis using digital occlusal device (occluscan).

The evaluation periods will be done at time of insertion (T0),6 month (T1),12 month(T2) and 18 month(T3) after framework insertion.

DETAILED DESCRIPTION:
thirty completely edentulous patients will be selected for the study from the outpatient's clinic of Prosthodontic Department, Faculty of Dentistry, Mansoura University.

The patients will be selected according to the following criteria:

1. lack of satisfaction of mandibular conventional dentures due to denture instability.
2. Atrophy of mandibular ridges with insufficient bone.
3. They were healthy, free from any systemic diseases relating to bone resorption.
4. All patients have sufficient inter-arch space >15 mm.
5. Maxillary and mandibular residual alveolar ridges covered by healthy non-inflamed mucosa with even compressibility.
6. Normal maxilla-mandibular relationship (class I Angle's classification).
7. All patients will have mandibular bone height not less than 8-10mm as verified by cone beam CT.
8. Sufficient inter-arch space not less than 23 mm as verified by tentative jaw relation. And restorative space not less than14 mm as verified by putty index technique.

Exclusion criteria included:

1- Systemic disorders affecting bone (such as uncontrolled diabetes mellitus and osteoporosis).

2- Local or general contraindication for surgical procedures. 3- History of chemotherapy or radiation therapy to the head and neck area. 4- Habits as heavy smoking and alcoholism. 5- Patients with T.M.J disorders or poor neuromuscular co-ordination.

1. For all patient's conventional complete denture will be constructed and adjusted for insertion and delivery.
2. A cone beam C.T will be done for each patient to determine the bone quality and quantity.
3. A surgical stent will be designed and fabricated to allow accurate implant placement of two axially placed anterior implants and two distally tilted posterior implants by about 30 degree to support mandibular overdenture.
4. Surgical placement of implant fixtures on its sites will be done.
5. Multiunit abutments were screwed to the distal implants.
6. The conventional mandibular denture will be modified to act as immediate fixed prosthesis that replace lost teeth and gingival tissues.
7. After three months, the Polyetheretherketone (PEEK) frame that connects the four implants will be constructed using digital scan and CAD CAM manufacturing.
8. The milled frame was fixed to the metal caps using DTK cement
9. The BioHPP framework will have prepared abutments projecting from it. After processing, the framework will be tried in patient mouth for passive fit.
10. Wax interocclusal record was made to establish the occlusal relationship with opposing teeth.

    According to the artificial teeth, the patients will be divided into two groups:
    * Group (I): PEEK framework veneered with nanocomposite resin(visio-lign)
    * Group (II): PEEK framework veneered with zirconia
11. The inner surface of the artificial teeth will be etched using hydrophosphoric acid then silane will be used and light cured resin cement will be used for cementation of the artificial teeth to the PEEK framework
12. The occlusal scheme used with the opposing maxillary denture will be lingualized balanced occlusion to enhance the stability of mandibular implant overdentures.

Methods of evaluation:

1- Occlusal force analysis using digital occlusal device (occluscan).

The evaluation periods will be done at time of insertion (T0), 6 month (T1), 12 month (T2) and 18 month (T3) after framework insertion.

ELIGIBILITY:
Inclusion Criteria:

* 1- lack of satisfaction of mandibular conventional dentures due to denture instability. 2- Atrophy of mandibular ridges with insufficient bone. 3- They were healthy, free from any systemic diseases relating to bone resorption. 4- All patients have sufficient inter-arch space >15 mm. 5- Maxillary and mandibular residual alveolar ridges covered by healthy non-inflamed mucosa with even compressibility. 6- Normal maxilla-mandibular relationship (class I Angle's classification). 7- All patients will have mandibular bone height not less than 8-10mm as verified by cone beam CT. 8- Sufficient inter-arch space not less than 23 mm as verified by tentative jaw relation. And restorative space not less than14 mm as verified by putty index technique.

Exclusion Criteria:

* 1- Systemic disorders affecting bone (such as uncontrolled diabetes mellitus and osteoporosis). 2- Local or general contraindication for surgical procedures. 3- History of chemotherapy or radiation therapy to the head and neck area. 4- Habits as heavy smoking and alcoholism. 5- Patients with T.M.J disorders or poor neuromuscular co-ordination.

Ages: 45 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2023-09-04 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
occlusal stability | The evaluation periods will be done at time of insertion (T0), 6 month (T1), 12 month (T2) and 18 month (T3) after framework insertion
  Occlusal stability using digital occlusal device (occlusense)

CONTACTS AND LOCATIONS:
Overall Officials: Mansoura U Faculty of dentistry, Principal Investigator — Mansoura University Faculty of Dentistry, Prosthodontics department
Locations (1):
- Mansoura University, Faculty of dentistry, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided